CLINICAL TRIAL: NCT02696889
Title: Autologous Stem Cell Therapy for Premature Ovarian Insufficiency and Low Ovarian Reserve
Brief Title: Rejuvenation of Premature Ovarian Failure With Stem Cells
Acronym: ROSE-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ayman Al-Hendy, Professor of Obstetrics and Gynecology, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0277
Record Dates: First submitted 2016-02-16; First posted 2016-03-02 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Primary Ovarian Insufficiency; Low Ovarian Reserve; Premature Ovarian Failure
Keywords: Infertility; Premature Ovarian Failure; Stem Cells; Amenorrhea; Low Ovarian Reserve; Ovarian Insufficiency; Premature menopause; Premature Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility; Amenorrhea; Menopause, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ROSE-1 Protocol (Experimental): Patients with POF, POI or Low Ovarian Reserve choosing to enroll will be provided informed consent for Rejuvenation of Premature Ovarian Failure With Stem Cells (ROSE-1). They will undergo diagnosis and screening confirming diagnosis including History and Physical Exams, Labs and Diagnostic Procedures. Following final approval and under anesthesia, bone marrow aspiration with separation of the bone marrow derived stem cell fraction will be performed. Diagnostic laparoscopy will allow for assessment of pelvic anatomy and subsequent injection of the bone marrow derived stem cells into the right ovary.
  Interventions: Procedure: ROSE-1 Protocol

INTERVENTIONS:
Procedure: ROSE-1 Protocol — A bone marrow aspiration will be performed under anesthesia in preparation for a diagnostic laparoscopy for full evaluation of the pelvic anatomy. Following laparoscopy, injection of BMSCs into the right ovary will occur.

SUMMARY:
The ROSE-1 study is designed to determine the efficacy of bone marrow derived stem cell therapy on ovarian function recovery in subjects with idiopathic and other types of premature or primary ovarian failure (POF or POI) and low ovarian reserves.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI), formerly referred to as premature ovarian failure (POF), is defined as hypergonadotropic ovarian insufficiency occurring prior to age 40 (1). It is surprisingly common and affects approximately 1% of women below the age of 40 (2, 3). The incidence is 10% to 28% in women with primary amenorrhea and 4% to 18% in women with secondary amenorrhea (2). The clinical manifestations include amenorrhea and abnormally high levels of luteinizing (LH) and follicle stimulating hormone (FSH) and low levels of Anti Mullerian Hormone (AMH). The etiology of POI is unknown in most cases. It can be caused by a combination of inherited conditions such as immune disorders, environmental toxins and iatrogenic injury (2, 3). The majority of patients with POI are considered to have idiopathic premature ovarian insufficiency because usually no cause can be identified (3). POI has been shown to be associated with an increased incidence of other conditions, including Alzheimer's, cardiovascular and immune system diseases, metabolic syndrome, osteoporosis, diabetes and cancer of reproductive organs. POI is characterized by loss of secondary follicles, arrested folliculogenesis, decreased estrogen production, and infertility (3). The mechanism of ovarian insufficiency is most likely accelerated follicular atresia but detailed pathogenesis is yet to be fully understood (2).

In women younger than 40, at least two menopausal FSH levels (≥40 IU/L) will be sufficient for the diagnosis of POI. It is not essential to have amenorrhea for the diagnosis of POI. Subjects with oligomenorrhea or low ovarian reserve and elevated FSH, referred to as transitional ovarian insufficiency (TOI), or at least 4 months amenorrhea together with FSH levels exceeding 40 IU/liter, and are included in this category. Spontaneous menstrual cycles can sometimes be seen after the diagnosis of POI as well. Resumption of normal ovarian function, albeit temporary, in patients with normal karyotypes has been documented in 10 to 20% of patients; thus, spontaneous resumption of fertility is possible (1).

No therapeutic intervention has proven effective in restoring fertility in patients with POI. Currently, egg donation remains the only reliable method to establish a pregnancy in women with POI (2, 3). Even though this approach is attainable, resulting children will not be genetically related to the recipient mother. Furthermore, egg donation is not ethically acceptable to many couples. Various attempts at ovarian stimulation patients with POI are usually unsuccessful because they are poor responders. Therefore, the diagnosis of POI can cause great physical and mental suffering among these patients. Thus, there is critical need to develop novel effective approaches for the treatment of POI.

Throughout life, there is an ongoing physiological level of atresia of oocytes. A decreased germ cell endowment combined with an increased rate of germ cell destruction can explain POI (1). The current concept that the ovary has a static ovarian reserve is entirely at odds with the germ cell dynamics. Current research supports the concept that the ovary continues to produce new germ cells into adult life, however, whether this occurs in humans is not universally accepted. Recent research suggests that diminished ovarian reserve is a result of the aging of the niche rather than a defect in the germ cells (4-6). Anti-mullerian hormone has been used as a reliable biomarker for ovarian reserve in humans and the circulating AMH levels change with age as follows:

20-25: 1.23-11.51 ng/mL 26-30: 1.03-11.10 ng/mL 31-35: 0.66-8.75 ng/mL 36-40: 0.42-8.34 ng/mL 41-46: 0.26-5.81 ng/mL 47-54: <0.82 ng/mL Emerging evidence suggests that bone marrow-derived mesenchymal stem cells (BMSCs) could restore the structure and function of injured tissues (7). During embryologic development, cells of the mesodermal layer give rise to multiple mesenchymal tissue types including bone, cartilage, tendon, muscle, and fat and marrow stroma (8). These precursor cells, also present in the postnatal organism, are referred to as mesenchymal stem cells. These stem cells have been shown to retain their developmental potential following extensive sub-cultivation in vitro. Implantation of culture-expanded mesenchymal stem cells has been demonstrated to effect tissue regeneration in a variety of animal models and depends on local factors to stimulate differentiation into the appropriate phenotype (8).

Recent studies suggest that stem cell therapy holds promise in treatment of variety of diseases including reproductive dysfunction. In a recent investigation by Ghadami et al (2012) in our lab at Augusta University in Georgia, BMSC treated animals resumed ovarian function (9). In another investigation by Lui et al (2014), granulosa cell apoptosis induced by cisplatin was reduced when BMSCs were migrated to granulosa cells in vitro. In this study, chemotherapy-induced POI rats were injected with BMSCs. The BMSCs treatment group's antral follicle count and estradiol levels increased after 30 days, compared with untreated POI group (10). In a recent clinical trial in Egypt, Edessy et al (2014) evaluated the therapeutic potential of autologous mesenchymal bone marrow stem cells transplantation in women with POI. Ten patients with POI were selected and their ovaries were injected with autologous BMSC at time of laparoscopy. The results revealed resumption of menstruation in one case after 3 months; two cases showed focal secretory changes after having atrophic endometrium (11). According to these results, BMSC seem to have the ability to revive prematurely failed ovaries both in their hormonal and follicular development abilities.

Furthermore, in this clinical trial, while at Augusta University, Georgia, USA, we have successfully initiated two cases so far (8/10/2017). Both patients have tolerated the procedure very well with no reported side effects or complications. Our first patient resumed menses after 6 months post stem cell injection and she demonstrated decreasing levels of serum FSH and increasing serum Estradiol levels (from undetectable levels pre-procedure, as well as the one week, one month and 3 months' time points assessments to 96pg/ml at the 6 months' time point (latest data available so far). She also reported amelioration of her post-menopausal symptoms including a decrease in hot flashes frequency and severity, decreased vaginal dryness and improved sleeping patterns. The second patient will be finished with the post-procedure follow up period on 2/21/2018.

Stem cell therapy has been shown to be beneficial and effective in various disease processes. The safety of the stem cell therapy has been assessed in multiple clinical trials. Although, autologous mesenchymal stem cell therapy for premature ovarian insufficiency is a novel approach, the safety and success of such stem cell therapy has been demonstrated in many other disease processes including graft versus host disease, acute myocardial infarction, acute respiratory distress syndrome (ARDS) and many other diseases (12-14). There are additional ongoing trials (Pilot -Phase III) to further assess risk and safety of stem cell based therapies (15-17). This interventional pilot clinical study will investigate the use of stem cell therapy to restore steroidogenesis, folliculogenesis, menstruation, and fertility in participants.

ELIGIBILITY:
Inclusion Criteria

* Able to understand and communicate in English language
* Signed and dated informed consent
* Female over the age of 18
* Diagnosis of premature ovarian insufficiency: At least two menopausal FSH levels (≥ 40 IU/L) and/or Primary or secondary amenorrhea at least for 3-6 months OR Diagnosis of low ovarian reserve defined as: AMH < _0.42 ng/ML & FSH >20 IU/L, and/or failure of prior attempts of assisted reproductive techniques due to limited ovarian response (poor responder).
* Normal karyotype 46, XX.
* Presence of at least one ovary
* Acceptable uterine anatomy (by any clinically and/or imaging acceptable methods)
* Normal thyroid function as evidence by normal serum Thyroid Stimulating Hormone (TSH) levels.
* Agree to report any pregnancy to the research staff immediately.
* Willing and able to comply with study requirements and follow up instructions.
* No other causes of female infertility in the subject

If subject is planning to pursue pregnancy: Presence of at least unilateral tubal patency (with any clinically acceptable methods).

Exclusion Criteria

* Unable to understand and communicate in English language
* Currently pregnant or breast-feeding
* Has a history of, or evidence of current gynecologic malignancy within the past three years
* Presence of adnexal masses indicating the need for further evaluation
* Major mental health disorder that precludes participation in the study
* Active substance abuse or dependence
* Unfit or unwilling to undergo laparoscopy; has contraindication to laparoscopic surgery and/or general anesthesia
* Current or recent (within the past 2 weeks) use of the following medications: Oral or systemic corticosteroids, Hormones (estrogen, progestins, oral contraceptives), Danazol, anticoagulants, herbal or botanical supplements with possible hormonal effects. Washout will be allowed.
* Medical conditions that are contraindicated in pregnancy
* Type I or Type II diabetes mellitus, or if receiving antidiabetic medications
* Known significant anemia (Hemoglobin <8 g/dL).
* Untreated deep venous thrombosis, and/or pulmonary embolus
* Untreated cerebrovascular disease
* Known heart disease (New York Heart Association Class II or higher).
* Known Liver disease (defined as Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)>2 times normal, or total bilirubin >2.5 mg/dL).
* Known Renal disease (defined as Blood urea nitrogen (BUN)>30 mg/dL or serum creatinine > 1.6 mg/dL).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02-06 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Improved diagnostic hormonal levels | 18 months
  Reduction of 50% in FSH values; increase in AMH and Estradiol levels (30%)

SECONDARY OUTCOMES:
Resumption of menses | 18 months
  Resumption of menses. Improved quality of life using the North American Menopausal Society (NAMS) validated menopause health questionnaire.
Improved clinical hormone levels | 18 months
  Improvement in hormonal levels toward normal ranges. Hormones may include FSH/LH; Estradiol/ progesterone;Inhibin; Anti- Mullerian Hormone
Achievement of pregnancy | 18 months
  Achievement of pregnancy by natural or assisted conception methods as may be deemed appropriate by the patient and her primary provider.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Al-Hendy, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Igboeli P, El Andaloussi A, Sheikh U, Takala H, ElSharoud A, McHugh A, Gavrilova-Jordan L, Levy S, Al-Hendy A. Intraovarian injection of autologous human mesenchymal stem cells increases estrogen production and reduces menopausal symptoms in women with premature ovarian failure: two case reports and a review of the literature. J Med Case Rep. 2020 Jul 18;14(1):108. doi: 10.1186/s13256-020-02426-5. PMID 32680541